CLINICAL TRIAL: NCT06011148
Title: Clinical Data Collection on Perceval S Sutureless Prosthetic Aortic Valve in the Chinese Population
Status: Not yet recruiting | Type: Observational
Sponsor: Corcym S.r.l (Industry)
Responsible Party: Sponsor
Other Study IDs: CCH803
Record Dates: First submitted 2023-08-01; First posted 2023-08-25 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Aortic Valve Disease
MeSH Terms: conditions — Aortic Valve Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Subject implanted with Perceval S sutureless prosthetic heart valve: Subjects who have been implanted with Perceval S sutureless prosthetic heart valve from 2022 onward and subjects that will be implanted up to study closure.
  Interventions: Device: Perceval S sutureless heart valve

INTERVENTIONS:
Device: Perceval S sutureless heart valve — Aortic Valve Replacement with Perceval S sutureless heart valve

SUMMARY:
The objective of the study is to evaluate the safety information on the Perceval S sutureless prosthetic heart valve after the implantation for aortic valve disease.

The study is designed as a post-market, observational, non-interventional retrospective and prospective registry.

DETAILED DESCRIPTION:
In order to monitor the ongoing safety of the Perceval S as part of regulatory requirements, the study aims to retrospectively collect safety outcomes and performance data in patients with aortic valve disease implanted with Perceval S since 2022. The data will be used for regulatory purposes, to support the re-certification of the valve in the Chinese market.

Serious Adverse Events (SAEs) such as valve-related death, structural valve deterioration, cerebral thromboembolism, stroke, Transient Ischemic Attack, non-cerebral thromboembolism, major bleeding, re-operation will be studied to describe the safety profile of the valve.

Hemodynamic data from site reported echocardiography finding (mean gradient, peak gradient, effective orifice area, effective orifice area indexed, incidence and degree of PVL and central leak) at hospital discharge will also be evaluated. Data of approximately 80 subjects will be collected in four clinical sites in China.

ELIGIBILITY:
Inclusion Criteria:

1. Subject who has been implanted with Perceval S sutureless aortic heart valve
2. Subject (legal representative or family member) who has signed the approved informed consent or would provide verbal informed consent/ signed and dated informed consent, and available medical information

Exclusion Criteria:

1. Subject (legal representative or family member) who do not provide consent to the data collection

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects who have been implanted with Perceval S sutureless prosthetic heart valve from 2022 onward and subjects that will be implanted up to study closure.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Mortality | up to 1 year
  The number and percentage of subjects died
Structural valve deterioration | up to 1 year
  The number and percentage of subjects with Structural valve deterioration
Cerebral thromboembolism | up to 1 year
  The number and percentage of subjects with Cerebral thromboembolism
Stroke | up to 1 year
  The number and percentage of subjects with stroke
Transient Ischemic Attack (TIA) | up to 1 year
  The number and percentage of subjects with Transient Ischemic Attack (TIA)
Non-cerebral thromboembolism | up to 1 year
  The number and percentage of subjects with non-cerebral thromboembolism
Major bleeding | up to 1 year
  The number and percentage of subjects with major bleeding
Re-operation | up to 1 year
  The number and percentage of subjects with re-operation

SECONDARY OUTCOMES:
Aortic Mean Pressure Gradient (MPG) | at discharge or 7 days post-procedure (whichever comes first)
  Decrease of MPG from baseline
Aortic Peak Pressure Gradient (PPG) | at discharge or 7 days post-procedure (whichever comes first)
  Decrease of PPG from baseline
Effective Orifice Area (EOA) | at discharge or 7 days post-procedure (whichever comes first)
  Increase of EOA from baseline
Effective Orifice Area Index (EOAi) | at discharge or 7 days post-procedure (whichever comes first)
  Increase of EOAi from baseline
Aortic Regurgitation | at discharge or 7 days post-procedure (whichever comes first),
  incidence and degree of paravalvular and central leak

CONTACTS AND LOCATIONS:
Overall Officials: Sara Gaggianesi, Study Director — Corcym S.r.l